CLINICAL TRIAL: NCT00917592
Title: Prospective Randomized Clinical Trial Assessing the Efficacy of a Short Course of Intravenous Amoxicillin Plus Clavulanic Acid Followed by Oral Antibiotic in Patients With Uncomplicated Acute Diverticulitis
Brief Title: Trial Assessing the Efficacy of a Short Course of Intravenous Antibiotic Followed by Oral Antibiotic in Uncomplicated Acute Diverticulitis
Acronym: DANC-05
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Consorci Sanitari de Terrassa (Other)
Collaborators: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Yolanda Ribas, Principal Investigator, Consorci Sanitari de Terrassa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DANC-05
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Diverticulitis
Keywords: Diverticulitis
MeSH Terms: conditions — Diverticulitis | interventions — Amoxicillin; Clavulanic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Short intravenous amoxicillin plus clavulanic acid (Experimental): Intravenous antibiotic 48 hours followed by oral antibiotic for 10 days
  Interventions: Drug: amoxicillin plus clavulanic acid
- Long intravenous amoxicillin plus clavulanic acid (Active Comparator): Intravenous antibiotic for 7 days followed by oral antibiotic for 5 days
  Interventions: Drug: amoxicillin plus clavulanic acid

INTERVENTIONS:
Drug: amoxicillin plus clavulanic acid — intravenous amoxicillin plus clavulanic acid 1 gr every 8 hours 48 hours followed by oral amoxicillin plus clavulanic acid 1 gr every 8 hours for 10 days
Drug: amoxicillin plus clavulanic acid — intravenous amoxicillin plus clavulanic acid for 7 days followed by oral antibiotic for 5 days

SUMMARY:
Medical treatment of uncomplicated acute diverticulitis is not standardized and there is an enormous diversity in clinical practice. The investigators' aim was to demonstrate that uncomplicated diverticulitis can be managed with oral amoxicillin plus clavulanic acid with a short hospital admission.

DETAILED DESCRIPTION:
A prospective randomized trial was established to compare patients with uncomplicated diverticulitis who received oral antibiotic after a short course of intravenous antibiotic, with those who received intravenous antibiotic for a longer period. We included 50 patients, 25 in each group. Patients in group 1 begun oral antibiotic as soon as they improved and were discharged the day after. Patients in group 2 received intravenous antibiotic for 7 days. Both groups received oral antibiotic at discharge. The endpoint of the study was "failure of treatment" which was defined as the impossibility of discharging on the expected day, emergency admission or hospital readmission.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of uncomplicated acute diverticulitis confirmed by a computed tomography (CT) scan within 24-48 hours

Exclusion Criteria (prerandomization):

* immunocompromised patients
* pregnant women
* clinical suspicion or CT confirmation of complicated acute diverticulitis
* Karnofsky performance score less than 50%
* allergy to penicillin

Exclusion Criteria (postrandomization):

* withdrawal of the trial
* CT confirmation of complicated acute diverticulitis
* CT not conforming to acute diverticulitis
* CT performed 72 hours after the admission
* adverse reaction to the antibiotic
* bacteriemia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-12; Primary Completion 2008-05 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
failure of treatment | the 4th day (group 1) or the 8th day (group 2)

SECONDARY OUTCOMES:
emergency admission or hospital readmission for reasons related to the previous diverticulitis | 30 days after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Yolanda Ribas, MD, PhD, Principal Investigator — Consorci Sanitari de Terrassa
Locations (1):
- Consorci Sanitari de Terrassa, Terrassa, Barcelona, Spain